CLINICAL TRIAL: NCT05700760
Title: The ROSE Scale-up Study: Informing a Decision About ROSE as Universal Postpartum Depression Prevention
Brief Title: The ROSE Scale-up Study: Informing a Decision About ROSE as Universal PPD Prevention
Acronym: ROSES-II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Pacific Institute for Research and Evaluation (Other); Henry Ford Health System (Other); Butler Hospital (Other)
Responsible Party: Principal Investigator, Jennifer E. Johnson, C. S. Mott Endowed Professor of Public Health, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01MH130948 (NIH); STUDY00007607 (Other: MSU IRB Study ID)
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Postpartum Depression
Keywords: postpartum depression; antenatal depression; depression; prevention; depression prevention; pregnancy
MeSH Terms: conditions — Depression, Postpartum; Depression

STUDY DESIGN:
Intervention Model Description: ROSE vs Enhanced Care as Usual (CAU)
Who Masked: Outcomes Assessor
Masking Description: Research assistants will randomize participants to a study arm. The participant will be assigned to a new research assistant for the follow-up assessment, who is masked from the study arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ROSE (Reach Out, Stay Strong, Essentials for mothers of newborns) (Experimental): Evidence-based 5 session psychosocial intervention that has been found to prevent ~50% of postpartum depression among low-income, at risk women.
  Interventions: Behavioral: ROSE (Reach Out, Stay Strong, Essentials for mothers of newborns)
- Enhanced Care as Usual (CAU) (Active Comparator): Usual care at the study site does not include postpartum depression prevention. Instead, HFHS clinics try to screen for PPD that has already occurred and refer women for mental health care. Screening for existing PPD at these clinics primarily relies on the EPDS (10+), Perinatal women who score 10+ on the EPDS are referred for mental health services. Services received depends on follow-up, severity, and the mental health wait list. Our study will exclude women meeting criteria for likely current major depressive episode at baseline and assist them in obtaining mental health care. Enhanced CAU consists of usual care + monitoring and emergency referral, as is required to fulfill ethical obligations to trial participants.
  Interventions: Behavioral: Enhanced Care as Usual (CAU)

INTERVENTIONS:
Behavioral: ROSE (Reach Out, Stay Strong, Essentials for mothers of newborns) — Evidence-based 5 session psychosocial intervention that has been found to prevent ~50% of postpartum depression among low-income, at risk women.
  Arms: ROSE (Reach Out, Stay Strong, Essentials for mothers of newborns)
Behavioral: Enhanced Care as Usual (CAU) — Usual care at the study site does not include postpartum depression prevention. Instead, HFHS clinics try to screen for PPD that has already occurred and refer women for mental health care. Screening for existing PPD at these clinics primarily relies on the EPDS (10+), Perinatal women who score 10+ on the EPDS are referred for mental health services. Services received depends on follow-up, severity, and the mental health wait list. Our study will exclude women meeting criteria for likely current major depressive episode at baseline and assist them in obtaining mental health care. Enhanced CAU consists of usual care + monitoring and emergency referral, as is required to fulfill ethical obligations to trial participants.
  Arms: Enhanced Care as Usual (CAU)

SUMMARY:
The Reach Out, Stand Strong, Essentials for New Mothers (ROSE) program is an evidence-based intervention that prevents half of cases of postpartum depression and was one of two interventions recommended by the US Preventive Services Task Force in 2019. All effectiveness trials of ROSE and of the other recommended PPD prevention intervention included only low-income women a single risk factor that doubles incidence of PPD. Thus, the existing evidence base for PPD prevention consists primarily of women at increased risk for PPD. Based on data from the PIs' current implementation study of ROSE, many healthcare and community agencies in this implementation trial (78%) find it is more feasible for them to provide or offer ROSE to every woman as part of their standard workflow, than it is to create a screening and referral process for at risk women. In addition to being more feasible for agencies, universal prevention may also be advantageous because the cost of a screening false negative (resulting in a preventable case of PPD; $32,000) far exceeds the cost of ROSE delivery ($50-$300/woman). Effectiveness of ROSE among low-income women at risk for PPD is known (ROSE prevents ~50% of PPD cases). To inform a recommendation about using ROSE as universal vs. selective or indicated prevention, we need to determine the effectiveness of ROSE among general populations of women, including women screening negative for PPD risk. Thus, this project will assess ROSE effectiveness across PPD risk levels and across prevention approaches in a sample of 2,320 women from a large regional health system (based in Detroit, MI). Each proposed aim gathers a piece of information missing that is needed to guide decision-making about ROSE as universal prevention. We will assess ROSE as universal, selective, and indicated prevention in terms of: (1) ROSE effectiveness relative to a control for each prevention approach in preventing PPD and improving functioning; (2) cost outcome, (3) equity and (4) scalability of each prevention approach; and (5) mechanisms of ROSE effects across PPD risk levels. We will integrate results to advise about ROSE as universal prevention. This definitive PPD prevention trial will show how best to get an evidence-based program to those who need it in settings where they receive perinatal care by addressing a pragmatic and novel question (should ROSE be universal prevention?) and by examining equity and cost-outcome of universal vs. other prevention approaches.

DETAILED DESCRIPTION:
In 2019, the US Preventive Services Task Force (USPSTF) issued a recommendation indicating that it is possible to prevent postpartum depression through counseling interventions. The Reach Out, Stand Strong, Essentials for New Mothers (ROSE) program was one of the two interventions mentioned by name serving as a basis for the recommendation. ROSE was tested in 4 randomized trials in community prenatal settings with racially/ethnically diverse low-income adult pregnant women and prevented ~50% postpartum depression (PPD) cases. ROSE is scalable in that: (1) it does not require mental health clinicians or licensed providers of any kind; (2) it has a flexible delivery structure (e.g., group vs. individual, timing during pregnancy); (3) it is the shorter (5 vs. 8-17 sessions) of the two interventions described in the USPSTF report. PIs Johnson and Zlotnick (the developer of ROSE) are in Year 4 of an implementation trial examining how much technical support is needed for various kinds of agencies to implement and sustain ROSE over time (R01 MH114883). That trial enrolled 98 agencies serving low income women nationally (i.e., settings where women receive perinatal care), including prenatal clinics, home visiting, Healthy Start, and doula groups, among others. It answers many of the questions posed in this RFA, including identifying: (1) a "service-ready efficacious preventive intervention" that is "scalable and can be delivered with fidelity by setting providers;" (2) "strategies to train providers and support delivery of evidence-based approaches with fidelity across health care and community settings;" (3) implementation barriers and facilitators; and (4) effective implementation strategies. However, that trial raised a question about the USPSTF recommendation.

Universal vs. selective or indicated prevention. All effectiveness trials of ROSE and of the other recommended PPD prevention intervention included only low-income women, a single risk factor that doubles incidence of PPD. Three of the 4 ROSE trials included women who were screened for additional risk for PPD per the Cooper survey to maximize trial power. Because the existing evidence base consisted of women at increased risk for PPD, the USPSTF recommendation suggested that "clinicians provide or refer… persons who are at increased risk of perinatal depression to counseling interventions," and called for "more studies on the use of tools for risk assessment." However, most of the healthcare and community agencies in our implementation trial (78%) provide or offer ROSE to every woman as part of their standard work flow (i.e., provide it as universal prevention), finding this more feasible than creating a screening and referral process for indicated or selective prevention. Most of the other agencies use provider judgment to refer to ROSE. Only 7% use a screening tool (typically the Edinburgh) for ROSE referral. In addition to being more feasible, universal prevention may be better because: (1) the cost of a screening false negative (resulting in a preventable case of PPD; $32,000) far exceeds the cost of ROSE delivery ($50-300/woman); (2) women who already face societal stigma (racial/ethnic minorities, undocumented) can be fearful about consequences and feel further stigmatized when a screener singles them out as needing PPD prevention. This project assesses effectiveness, cost-outcome, equity, and scalability of using ROSE as universal vs. selective or indicated prevention for PPD using commonly available/existing screening tools. We expect universal prevention to be optimal. Effectiveness of ROSE among low-income women at risk for PPD is known (ROSE prevents ~50% of PPD cases). To inform a recommendation about using ROSE as universal vs. selective or indicated prevention, we need to determine the effectiveness of ROSE among all pregnant persons, including those screening negative for PPD risk (defined in various ways; Section A6). We will enroll 2,320 people receiving prenatal care in a large regional health system (based in Detroit, MI), assess them with PPD risk tools (chosen for ease of use, wide use, or availability in electronic health records), randomize everyone to ROSE or to enhanced care as usual (ECAU), and collect information needed to inform a decision about ROSE as universal PPD prevention. Each proposed aim gathers a piece of information missing in the USPSTF report to guide decision-making. We will assess ROSE as universal, selective, and indicated prevention in terms of:

1. ROSE effectiveness relative to ECAU for each prevention approach for (i) SCID5 major depressive episode (primary) and (ii) functioning in the 6 months after birth. We will explore effects between baseline and birth.
2. Cost-outcome comparison of universal vs. selective or indicated prevention in terms of PPD and functioning. Because it prevents costly false negatives, universal prevention is almost always cost-beneficial.
3. Equity: (a) Percent false negative screens for minority vs. non-Hispanic white women; (b) minority status as a moderator of outcome across risk levels; (c) PPD cases that would be prevented by ROSE as universal prevention that would not be prevented under selective/indicated for minority vs. non-Hispanic white women.
4. Scalability as indicated by: (a) cost-outcome comparison of universal vs. indicated prevention (Aim 2); (b) a scalability measure and qualitative interviews with the 98 agencies in the past ROSE implementation trial about how they decided on universal vs. some other kind of prevention and how it went in their settings.
5. Mechanisms of ROSE effects across PPD risk levels. We will integrate results to advise about ROSE as universal prevention. This study fits the RFA by assessing how best to get an evidence-based program to those who need it in settings where they receive perinatal care, by addressing a pragmatic and novel question (should ROSE be universal prevention?), and by examining equity.

B. Innovation B1. This will be the first fully-powered RCT to assess universal vs. selective or indicated prevention of an evidence-based intervention for PPD in terms of prevention of PPD cases. The USPSTF recommendation on prevention of postpartum depression (i.e., that "clinicians provide or refer pregnant and postpartum women who are at increased risk of perinatal depression to counseling interventions") is new (2019) and was limited to women at elevated risk for PPD because that is what the evidence to date consisted of (i.e., trials among women at elevated risk for PPD). However, our current 98-agency implementation trial and other factors suggest that universal prevention may be more scalable, cost-effective, and equitable than selective or indicated prevention for PPD. This trial will be the first to examine the advisability of universal vs. selective or indicated PPD prevention (a) at all, & (b) with respect to equity, scalability, and comparative cost.

B2. This definitive trial will be the largest PPD prevention trial to date. Among other advantages, this provides better power than previous studies to examine race/ethnicity by intervention interactions.

B3. This trial will be the first to explore ROSE as antenatal depression (AD) prevention.

B4. EPDS as a predictor of future PPD. The EPDS is a well-validated and almost ubiquitously used measure of perinatal depressive symptoms and it makes sense that elevated symptoms likely predict future disorder. However, no previous study has ever tested the EPDS as a predictor of future development of full PPD (only its correlation with current disorder), despite being used this way in clinical practice. A bonus additional feature of this trial is that we can use the control condition (n~1,160) to evaluate the predictive validity of this commonly used measure. Currently, no AD symptom measure has been validated as a predictor of PPD.

B5. Scalability is a relatively understudied area of implementation science. This study will provide the first (quantitative and qualitative) analysis of scalability of universal, selective, and indicated PPD prevention.

Approach: Research Design This project informs use of ROSE as universal vs. selective or indicated prevention for PPD by assessing: (1) ROSE effectiveness for each prevention approach among 2,320 women in terms of (i) SCID5 major depressive episode in the 6 months after birth (primary), and (ii) functioning. (2) Cost-outcome comparison of universal vs. selective or indicated prevention in terms of PPD and functioning (equation in Section D2.11). Savings from preventing false negatives (PPD cases among "low risk" women) drives this comparison. (3) Equity: (a) percent false negative screens for minority vs. non-Hispanic white women; (b) minority status as a moderator of outcome across risk levels; (c) PPD cases that would be prevented by ROSE as universal prevention that would not be prevented under selective/indicated for minority vs. non-Hispanic white women. (4) Scalability of universal vs. other kinds of prevention as indicated by: (a) cost-outcome analyses (Aim 2); (b) a scalability measure and qualitative interviews with the 98 agencies in the ROSE implementation trial. (5) Mechanisms of ROSE effects across PPD risk levels.

ELIGIBILITY:
Inclusion Criteria:

1. Is aged 18 or older
2. Is receiving prenatal services within the U.S
3. Is between 12-32 weeks pregnant
4. Speaks and understand English well enough to understand questionnaires when they are read aloud
5. Has access to a telephone through owning one, a relative/friend, or an agency
6. Is willing and able to provide the name and contact information of at least two locator persons

Exclusion Criteria:

1. Has a current major depressive episode
2. Has current or past diagnosis of a bipolar disorder or a psychotic disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2320 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
SCID-5 Major Depressive Episode | through 6 months after birth
  The SCID is the gold standard diagnostic assessment of major depressive episode.

SECONDARY OUTCOMES:
SF-12 | Baseline (during pregnancy and 6 months after birth)
  Functioning will be measured using the SF-12, a brief, widely used measure of physical and mental health functioning that also provides our secondary cost-effectiveness measure.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E Johnson, PhD, Principal Investigator — Michigan State University; Caron Zlotnick, PhD, Principal Investigator — Butler Hospital
Locations (1):
- Michigan State University, Flint, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Participant data will be shared to the National Institute of Mental Health Data Archive (NDA).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data sharing will occur on NIH-designated timelines.
Access Criteria: Participant data will be shared to the National Institute of Mental Health Data Archive (NDA).

REFERENCES:
- [Derived] Johnson JE, Loree AM, Sikorskii A, Miller TR, Carravallah L, Taylor B, Zlotnick C. Study protocol for the ROSE Scale-Up Study: Informing a decision about ROSE as universal postpartum depression prevention. Contemp Clin Trials. 2023 Sep;132:107297. doi: 10.1016/j.cct.2023.107297. Epub 2023 Jul 18. PMID 37473848